CLINICAL TRIAL: NCT02343705
Title: Evaluation of the Latella Knee Implant System for Medial Osteoarthritis Pain Reduction (Latella-2 Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor election
Sponsor: Cotera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0001
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latella Knee Implant System (Experimental)
  Interventions: Device: Latella Knee Implant System

INTERVENTIONS:
Device: Latella Knee Implant System

SUMMARY:
The objective of the Latella-2 study is to demonstrate the safety and efficacy of the Latella Knee Implant System for the reduction of medial osteoarthritis knee pain.

ELIGIBILITY:
Inclusion Criteria:

* History of pain due to medial osteoarthritis
* Qualifying baseline pain scores
* Kellgren-Lawrence Grades 2-3

Exclusion Criteria:

* Osteoporosis
* Rheumatoid arthritis
* Joint instability
* Metal ion allergy
* Permanent implant in or around the knee joint
* Prior anterior cruciate ligament reconstruction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Efficacy assessed by KOOS pain score at 6 months after treatment with the Latella Implant | 6 Months
Primary Endpoint: Safety assessed by surgical re-intervention rate following implantation of the Latella device | 6 Months

SECONDARY OUTCOMES:
Changes in knee outcome measures (KOOS, IKDC, NRS) | 6, 12 and 24 months
Device and procedure complication rates | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Ramachandran, MD, Principal Investigator — Barts & The London NHS Trust
Locations (12):
- Netherlands (5):
  - Slotervaart Hospital, Amsterdam
  - Amphia Ziekenhuis, Breda
  - St. Anna Hospital, Geldrop
  - University Hospital Maastricht, Maastricht
  - Isala, Zwolle
- Spain (4):
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (3):
  - Royal London Hospital, London
  - Norfolk & Norwich University Hospital, Norwich
  - Morriston Hospital, Swansea